CLINICAL TRIAL: NCT03253757
Title: PrEP Impact Trial: A Pragmatic Health Technology Assessment of PrEP and Implementation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St Stephens Aids Trust (Other)
Collaborators: Public Health England (Other Government); NHS England (Other Government)
Responsible Party: Sponsor
Other Study IDs: SSCR104
Record Dates: First submitted 2017-06-16; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: HIV Infections
Keywords: PrEP; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This study is non-interventional. — This study is non-interventional.

SUMMARY:
HIV pre-exposure prophylaxis (PrEP) is the use of anti-HIV medicines by HIV negative people in order to prevent them from becoming HIV positive if exposed to HIV.

Currently, the combination drug containing tenofovir and emtricitabine is licensed in Europe for use as HIV PrEP. We know from previous studies worldwide that this combination drug is very good at reducing the risk of HIV infection and several countries have implemented PrEP programmes to provide PrEP to individuals at high risk of HIV.

However, it is difficult to effectively plan for a national PrEP programme in England without knowing how many people will need PrEP, how many will want to take PrEP, and how long they will stay on PrEP.

In order to find this out, the PrEP Impact Trial will make PrEP available to at least 10,000 people over three years. HIV negative men and women attending sexual health clinics in England will have their risk of HIV assessed by their care team and be offered PrEP if they meet the eligibility criteria. Through the trial we will be able to measure how many attendees at sexual health clinics meet eligibility criteria for PrEP, how many of these take up the offer of PrEP and how long they remain on PrEP for.

There will not be any additional tests other than those recommended for the safe delivery of PrEP. These include tests for sexually transmitted infections (STIs) and HIV as well as urine and blood tests to monitor kidney function. Information about attendances and test results will be anonymously collected through the existing data reporting system that sexual health clinics currently use to report to Public Health England.

ELIGIBILITY:
Inclusion Criteria:

The participant populations for this trial will be men and women attending GUM clinics who belong to one of three populations recognised to be at high risk for HIV, namely:

A. Men (cisgender and transgender) and transgender women who:

1. Have sex with men
2. Have had an HIV negative test during an earlier episode of care in the preceding year
3. Report condomless intercourse in the previous 3 months
4. Affirm their likelihood of having condomless intercourse in the next 3 months

B. HIV negative partners of an HIV positive person when:

1. The HIV positive partner is not known to be virally suppressed (<200 copies/ml for 6 months or more)
2. Condomless intercourse is anticipated before treatment of the HIV positive partner takes effect

C.HIV negative persons who:

1. Are clinically assessed and considered to be at similar high risk of HIV acquisition as those with a serodiscordant partner who is not known to be virally suppressed

Participants will therefore be considered eligible for trial enrolment if they fulfil all the following individual eligibility criteria:

1. Belongs to one of the three at high HIV risk populations described above
2. Aged 16 years or over (no upper limit)
3. Considered to be HIV negative on the day of enrolment
4. Willing and able to provide informed consent
5. Willing to adhere to the recommended PrEP regimen
6. Willing to re-attend the trial clinic at appropriate intervals for risk assessment

Exclusion Criteria:

1. An acute viral illness that could be due to HIV seroconversion
2. Any contraindication to Tenofovir Disoproxil (TD)/ Emtricitabine (FTC)-

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The participant populations for this trial will be men and women attending GUM clinics who belong to one of three populations recognised to be at high risk for HIV, namely:
  A. Men (cisgender and transgender) and transgender women who:
  1. Have sex with men
  2. Have had an HIV negative test during an earlier episode of care in the preceding year
  3. Report condomless intercourse in the previous 3 months
  4. Affirm their likelihood of having condomless intercourse in the next 3 months
  B. HIV negative partners of an HIV positive person when:
  1. The HIV positive partner is not known to be virally suppressed (<200 copies/ml for 6 months or more)
  2. Condomless intercourse is anticipated before treatment of the HIV positive partner takes effect
  C.HIV negative persons who:
  1. Are clinically assessed and considered to be at similar high risk of HIV acquisition as those with a serodiscordant partner who is not known to be virally suppressed
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
PrEP Eligibility | 3 years
  The proportion of GUM clinic attendees meeting the eligibility criteria for PrEP
PrEP Eligibility (duration) | 3 years
  The duration for which GUM clinic attendees are eligible for PreP
PrEP Uptake | 3 years
  The proportion of PrEP eligible GUM clinic attendees prescribed PrEP
PrEP Uptake (duration) | 3 years
  The duration for which eligible GUM clinic attendees use PrEP

SECONDARY OUTCOMES:
HIV | 3 years
  HIV diagnoses reported by sites and identified through the national surveillance dataset
STIs | 3 years
  STI diagnoses (gonorrhoea, chlamydia, syphilis and hepatitis C) reported in the national surveillance dataset
Adverse Events | 3 years
  1. Serious suspected adverse drug reactions reported using the yellow card system
  2. Antiretroviral resistance associated mutations in participants with incident HIV infection

IPD SHARING:
Plan to Share IPD: No
All data used in the study will be pseudo-anonymised and used for the purposes of determining the implementation of PrEP in England.

REFERENCES:
- [Derived] Sullivan AK, Saunders J, Desai M, Cartier A, Mitchell HD, Jaffer S, Ogaz D, Chiavenna C, Charlett A, Diamente V, Golombek R, Manavi K, Priestley C, Waters LJ, Milinkovic A, McOwan A, Estcourt C, Sabin CA, Rodger A, Gold D, Gazzard BG, McCormack S, Gill ON; Impact Study Group. HIV pre-exposure prophylaxis and its implementation in the PrEP Impact Trial in England: a pragmatic health technology assessment. Lancet HIV. 2023 Dec;10(12):e790-e806. doi: 10.1016/S2352-3018(23)00256-4. PMID 38040478